CLINICAL TRIAL: NCT06536036
Title: A Single Center, Randomized, Open Label, Single Dose, Two-Period, Crossover Phase I Study to Evaluate the Effect of Food (high-fat/standard Meal) on the Pharmacokinetics of SIM0270 in Healthy Adult Subjects in China
Brief Title: Evaluate the Effects of Food on the Pharmacokinetics of SIM0270
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nanjing Zaiming Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIM0270-102
Record Dates: First submitted 2024-07-16; First posted 2024-08-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High-fat meal group（Group1） (Experimental): Eight subjects were enrolled and administered single dose of 60mg SIM0270 under fasting condition in the first cycle, and administered single dose of 60mg SIM0270 under high-fat diet condition in the second cycle.
  Interventions: Drug: SIM0270
- High-fat meal group（Group2） (Experimental): Eight subjects were enrolled and administered single dose of 60mg SIM0270 under high-fat diet condition in the first cycle, and administered single dose of 60mg SIM0270 under fasting condition in the second cycle.
  Interventions: Drug: SIM0270
- Standard meal group（Group3） (Experimental): Eight subjects were enrolled and administered single dose of 60mg SIM0270 under fasting condition in the first cycle, and administered single dose of 60mg SIM0270 under standard meal condition in the second cycle.
  Interventions: Drug: SIM0270
- Standard meal group（Group4） (Experimental): Eight subjects were enrolled and administered single dose of 60mg SIM0270 under standard meal condition in the first cycle, and administered single dose of 60mg SIM0270 under fasting condition in the second cycle.
  Interventions: Drug: SIM0270

INTERVENTIONS:
Drug: SIM0270 — Use according to the prescribed protocol

SUMMARY:
This is a randomized, open label, single dose, two-period, crossover trial phase I study.

The purpose of this study is to evaluate the food effect on the pharmacokinetics（PK） of SIM0270 after oral administration under fasted, standard meal, or high-fat diet conditions.

DETAILED DESCRIPTION:
Part A High Fat Meal Test:

Sixteen healthy adult subjects are planned to be enrolled and randomly assigned to different dosing sequence groups (Group 1 and Group 2) in a 1:1 ratio for a two-period crossover trial. The subjects administered a single dose of SIM0270 under fasted, or high-fat diet conditions.

Part B Standard Meal Test (optional part):

Sixteen healthy adult subjects are planned to be enrolled and randomly assigned to different dosing sequence groups (Group 3 and Group 4) in a 1:1 ratio for a two-period crossover trial. The subjects administered a single dose of SIM0270 under fasted, or standard meal conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study content, process, and potential risks of this trial, and voluntarily sign the informed consent.
2. Male and female subjects,age 18-65 years
3. Male subjects weigh ≥50 kg, female subjects weigh ≥45 kg; BMI ≥ 19 and ≤ 28kg/m^2.
4. Subjects of childbearing potential agree to take recognized effective contraceptive measures during the study period and within 6 months after the last dose of the investigational product, starting from signing the informed consent.

Exclusion Criteria:

1. Neurological/psychiatric, respiratory, cardiovascular, gastrointestinal, hematological and lymphatic, endocrine, skeletal-muscular disorders , hepatic or renal insufficiency, or any other disease or condition that may affect the results of the study or the safety of the subjects.
2. With dysphagia or any history of gastrointestinal diseases that affect drug absorption.
3. There are risk factors for apical torsion type ventricular tachycardia, or other clinically significant abnormalities determined by research doctors.
4. Have a history of active or latent tuberculosis.
5. History of malignant tumors. Excluding cervical carcinoma in situ, non melanoma skin cancer, or stage I uterine cancer (with a disease-free interval of at least 5 years) that have received appropriate treatment.
6. Investigator believe that any acute or chronic disease may limit the ability of participants to complete and/or participate in this clinical study.
7. Individuals who are allergic to the research drug or any component of the research drug, have a specific history of allergies, or have an allergic constitution
8. Have used hormone replacement therapy or selective estrogen modulators within the year prior to enrollment.
9. Have used oral antibiotics within 4 weeks before enrollment or intravenous antibiotics within 8 weeks.
10. Any medication/product known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, used or intended to be used within one month prior to enrollment.
11. Used any prescription drugs/products within 2 weeks prior to enrollment or any over-the-counter drugs within 1 week prior to enrollment.
12. Received CYP3A4 strong inhibitor or strong inducer medication within 2 weeks prior to administration after signing the informed consent form.
13. The results of laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function), physical examination, vital signs, 12 lead electrocardiogram examination, chest anteroposterior and lateral radiographs, and abdominal ultrasound examination were determined by the researchers to be abnormal and clinically significant.
14. Screening period (mean) or baseline electrocardiogram examination shows heart rate<60 or>100 and QTcF interval>450 ms.
15. Pregnant women with fertility test results are positive or pregnant or lactating women.
16. Those who are positive for hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus (HIV) antibody and treponema pallidum antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
PK parameters: Peak Plasma Concentration (Cmax) | Day1 to Day 37
  Comparison of PK parameters of SIM0270 single dose in Chinese healthy adult subjects under fasted/ high-fat diet conditions, or under fasted/ standard meal conditions.
PK parameters:Area under the plasma concentration versus time curve (AUC) | Day1 to Day 37
  Comparison of PK parameters of SIM0270 single dose in Chinese healthy adult subjects under fasted/ high-fat diet conditions, or under fasted/ standard meal conditions.
PK parameters: Half-life (t1/2) | Day1 to Day 37
  Comparison of PK parameters of SIM0270 single dose in Chinese healthy adult subjects under fasted/ high-fat diet conditions, or under fasted/ standard meal conditions.

SECONDARY OUTCOMES:
Adverse events | From signing ICF until 18 days after the last dose of medication
  The incidence and grading of adverse events, as well as abnormal indicators of vital signs, physical examination, electrocardiogram, and laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China